CLINICAL TRIAL: NCT04389853
Title: Ambulatory Tubeless Mini Percutaneous Nephrolithotomy Versus Retrograde Intrarenal Surgery in the Management of Nephrolithiasis: A Randomized Controlled Clinical Study
Brief Title: Mini-PNCL vs fURS in Management of Nephrolithiasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thunder Bay Regional Health Research Institute (Other)
Responsible Party: Principal Investigator, Hazem Elmansy, Urology Surgeon, Thunder Bay Regional Health Research Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RP-645
Record Dates: First submitted 2020-05-05; First posted 2020-05-15 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Nephrolithiasis; Kidney Stone
MeSH Terms: conditions — Nephrolithiasis; Kidney Calculi

STUDY DESIGN:
Intervention Model Description: Randomized Control Study comparing two standard of care treatments.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Flexible ureteroscopy (fURS) (Active Comparator): Retrograde intrarenal surgery (RIRS) has gained much popularity especially when the role of SWL, in management of LPS, has been significantly diminished in the few last years5. RIRS is dependent mainly on flexible ureteroscopy (fURS). fURS increases the quality and performance of upper urinary tract exploration, allowing for the treatment of the majority of stones at all sites. Moreover, it is associated with no risk of renal parenchymal injuries and a very low risk of bleeding.
  Interventions: Procedure: Flexible ureteroscopy
- Mini-percutaneous nephrolithotomy (mini-PCNL) (Active Comparator): PCNL has regained popularity thanks to the possibility of using reduced calibers and modern technology, which has reduced the complications without compromising the stone clearance, and more efficient intracorporeal lithotripter modalities. However, PCNL is still a challenging surgical technique and can be associated with significant complications that may compromise its efficacy. In the present time, we have available calibers ranging from 4.8 to 30 French. Many reports advocate that morbidity after PCNL may be reduced by recent modifications, such as mini-PCNL (miniperc). One meta-analysis of mini-PCNL and conventional PCNL demonstrated that mini-PCNL had a greater safety profile with similar stone free rates (SFRs)4
  Interventions: Procedure: Mini-percutaneous nephrolithotomy

INTERVENTIONS:
Procedure: Flexible ureteroscopy — Retograde intrarenal surgery (RIRS) has gained much popularity especially when the role of SWL, in management of LPS, has been significantly diminished in the few last years5. RIRS is dependent mainly on flexible ureteroscopy (fURS). fURS increases the quality and performance of upper urinary tract exploration, allowing for the treatment of the majority of stones at all sites. Moreover, it is associated with no risk of renal parenchymal injuries and a very low risk of bleeding.
  Arms: Flexible ureteroscopy (fURS)
Procedure: Mini-percutaneous nephrolithotomy — PCNL has regained popularity thanks to the possibility of using reduced calibers and modern technology, which has reduced the complications without compromising the stone clearance, and more efficient intracorporeal lithotripter modalities. However, PCNL is still a challenging surgical technique and can be associated with significant complications that may compromise its efficacy. In the present time, we have available calibers ranging from 4.8 to 30 French. Many reports advocate that morbidity after PCNL may be reduced by recent modifications, such as mini-PCNL (miniperc). One meta-analysis of mini-PCNL and conventional PCNL demonstrated that mini-PCNL had a greater safety profile with similar stone free rates (SFRs).
  Arms: Mini-percutaneous nephrolithotomy (mini-PCNL)

SUMMARY:
The prevalence of nephrolithiasis is increasing over the last two decades, and kidney stones is a recurrent disorder, with lifetime recurrence risks reported to be as high as 50%. One of the most challenging stones is the lower pole (LP) nephrolithiasis.

The standard management of lower pole stones (LPS), is still controversial especially for stones smaller than 20 mm, with retrograde intrarenal surgery (RIRS) and mini-PCNL (miniperc) both demonstrated to be safe and effective methods for treating LPS with a diameter of 1-2 cm.

Selecting the optimal modality for treating renal calculi is challenging, as both techniques may be associated with different patient benefits and risk profiles. Despite the evolution of mini-PCNL and fURS techniques into clinical practice, there is a lack of comparative clinical data assessing SFRs and complication rates.

To the investigators' knowledge, no previous studies have addressed the outcome of ambulatory tubeless miniperc as a same day procedure, which this study will look to assess. The investigators are planning to discharge all participants home the night of surgery, without admission or insertion of nephrostomy tube. This will decrease the morbidity of miniperc and encourage head-to-head comparison with fURS in a prospective randomized protocol.

DETAILED DESCRIPTION:
The prevalence of nephrolithiasis is increasing over the last two decades, and kidney stones is a recurrent disorder, with lifetime recurrence risks reported to be as high as 50%. One of the most challenging stones is the lower pole (LP) nephrolithiasis. This could be explained by its antigravity location, acute angle with the renal pelvis and the narrow angle of the infundibulum. Therefore, the optimal management of LP calculi continues to be a dilemma. The standard management of lower pole stones (LPS), is still controversial especially for stones smaller than 20 mm, with competing interventions possessing advantages and disadvantages. Treatment options include percutaneous nephrolithotomy (PCNL), retrograde intrarenal surgery (RIRS), or shockwave lithotripsy (SWL).

PCNL has regained popularity thanks to the possibility of using reduced calibers and modern technology, which has reduced the complications without compromising the stone clearance, and more efficient intracorporeal lithotripter modalities. However, PCNL is still a challenging surgical technique and can be associated with significant complications that may compromise its efficacy. In the present time, surgeons have available calibers ranging from 4.8 to 30 French. Many reports advocate that morbidity after PCNL may be reduced by recent modifications, such as mini-PCNL (miniperc). One meta-analysis of mini-PCNL and conventional PCNL demonstrated that mini-PCNL had a greater safety profile with similar stone free rates (SFRs).

Another alternative option is RIRS. RIRS has gained much popularity especially when the role of SWL, in management of LPS, has been significantly diminished in the few last years. RIRS is dependent mainly on flexible ureteroscopy (fURS). fURS increases the quality and performance of upper urinary tract exploration, allowing for the treatment of the majority of stones at all sites. Moreover, it is associated with no risk of renal parenchymal injuries and a very low risk of bleeding.

RIRS and miniperc are both safe and effective methods for treating LPS with a diameter of 1-2 cm. The SFRs were comparable at the first postoperative day (90.2% vs. 93.2%) and the second month postoperatively (93.8% vs. 95.1%), for RIRS and miniperc, respectively. However, miniperc was associated with significant longer hospital stay and higher hospitalization costs.

Therefore, selecting the optimal modality for treating renal calculi is challenging, as both techniques may be associated with different patient benefits and risk profiles. Despite the evolution of mini-PCNL and fURS techniques into clinical practice, there is a lack of comparative clinical data assessing SFRs and complication rates.

To the investigators' knowledge, no previous studies have addressed the outcome of ambulatory tubeless miniperc as a same day procedure, which this study will look to assess. The investigators are planning to discharge all participants home the night of surgery, without admission or insertion of nephrostomy tube. This should decrease the morbidity of miniperc and encourage head-to-head comparison with fURS in a prospective randomized protocol.

The investigators will attempt to address whether there is a difference in clinical outcome between ambulatory mini percutaneous nephrolithotomy and flexible ureteroscopy in the management of lower pole kidney stones?

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects over 18 years of age at the time of enrollment.
2. Patients referred with single kidney stones of 10-20 mm in its largest diameter, or multiple stones involving a single calyx.
3. Written informed consent to participate in the study
4. Ability to comply with the requirements of the study procedures

Exclusion Criteria:

1. Congenital anatomic anomalies of the kidney, ureters or bladder.
2. Previous ipsilateral renal surgery within past five years.
3. Patients with ipsilateral distal ureteral stones or stricture.
4. Stone size > 20 mL or multiple kidney stones in different calyces.
5. Previous SWL treatment for the same stone.
6. Patients presented with a previously inserted ipsilateral ureteral stent.
7. Participants with active urinary tract infection until appropriately treated
8. Uncorrected coagulopathy (anticoagulants or blood thinners which cannot be withheld before surgery).
9. Pregnancy or morbid obesity
10. Participants with preexisting conditions, which, in the opinion of the investigator, interfere with the conduct of the study.
11. Participants who are uncooperative or cannot follow instructions.
12. Participants who lack the capacity to provide free and informed written consent.
13. Patients with solitary kidney.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2020-10-05 (Actual); Primary Completion 2024-04-24 (Actual); Study Completion 2024-04-24 (Actual)

PRIMARY OUTCOMES:
Stone-free status | 1-day
  Operation success will be evaluated with a non-contrast computed tomography (CT) scan on the first post-operative day, as per standard of care. Presence or absence of kidney stones will be confirmed via CT scan
Stone-free status | 4-weeks post-op
  Operation success will be re-evaluated with a non-contrast computed tomography (CT) scan at 4-weeks post-operation, as per standard of care. Presence or absence of kidney stones will be confirmed via CT scan

SECONDARY OUTCOMES:
To compare safety measures | 4 weeks
  Adverse events including perioperative bleeding, operative time, fluoroscopy time, need for blood transfusion, stone composition, fragmentation type, ureteral stenting, and urinary tract infection will be recorded intra and post-op
To compare stone free status of single use vs reusable fURS | 1-day post-op
  Subgroup analysis comparing two types of fURS treatments. In this study, participants randomized to the fURS cohort may receive either single use or reusable fURS are their standard of care treatment. The investigators plan to conduct a subgroup analysis comparing stone-free status 1-day post-op using a standard of care non-contrast CT scan.
To compare stone free status of single use vs reusable fURS | 4-weeks post-op
  Subgroup analysis comparing two types of fURS treatments. In this study, participants randomized to the fURS cohort may receive either single use or reusable fURS are their standard of care treatment. The investigators plan to conduct a subgroup analysis comparing stone-free status 4-weeks post-op using a standard of care non-contrast CT scan.
Assess the postoperative pain between both techniques | 1-day post-op
  Post-surgical pain will be assessed using a Visual Analog Scale (VAS) questionnaire. This questionnaire consists of 1 question asking participants to choose a number from 0-10 describing their pain at the current moment. A lower score indicates less pain, while a higher score indicates a higher degree of pain. For example a score of 0 indicates "No Pain", while a score of 10 indicates "Unbearable Pain".
Assess the postoperative pain between both techniques | 4-weeks post-op
  Post-surgical pain will be assessed using a Visual Analog Scale (VAS) questionnaire. This questionnaire consists of 1 question asking participants to choose a number from 0-10 describing their pain at the current moment. A lower score indicates less pain, while a higher score indicates a higher degree of pain. For example a score of 0 indicates "No Pain", while a score of 10 indicates "Unbearable Pain".

CONTACTS AND LOCATIONS:
Overall Officials: Hazem Elmansy, MD, Principal Investigator — Thunder Bay Regional Health Sciences Centre
Locations (1):
- Thunder Bay Regional Health Sciences Centre/Thunder Bay Regional Health Research Institute, Thunder Bay, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
There are no plans to share participant data with other researchers. Findings may be presented locally, nationally, and internationally at conferences. Any data presented will be de-identified and grouped prior to use, as to protect participant confidentiality.